CLINICAL TRIAL: NCT02483481
Title: Using Ultrasound Elastography to Predict Development of Sinusoidal Obstruction Syndrome
Brief Title: Using Ultrasound Elastography to Predict Development of SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 15060244
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Sinusoidal Obstruction Syndrome; Complications of Bone Marrow Transplant
Keywords: sinusoidal obstruction syndrome; ultrasound elastography; bone marrow transplant
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Shear Wave Ultrasound Elastography (Other)
  Interventions: Diagnostic Test: shear wave ultrasound elastography

INTERVENTIONS:
Diagnostic Test: shear wave ultrasound elastography — shear wave ultrasound elastography

SUMMARY:
Sinusoidal obstruction syndrome (SOS) is a potentially fatal hepatic veno-occlusive disease-affecting children following bone marrow transplantation (BMT). SOS most likely develops secondary to sinusoidal endothelial damage and subsequent obstruction. The disease can be separated into mild, moderate, and severe forms; almost all patients diagnosed with severe SOS will die from this disease. Children with severe SOS suffer from multi-organ failure with signs and symptoms of portal hypertension (ascites, varices, edema), renal and respiratory failure . Although these children may be few and far between, the mere severity of the disease process and awful prognosis factors are valid reasons for more medical attention. SOS is usually diagnosed via clinical criteria and, despite available prophylaxis and treatment, children continue to die from this devastating disease.

Quantitative shear wave ultrasound elastography with acoustic force radiation imaging is an emerging technology that uses ultrasound pressure waves to provide an estimate of tissue stiffness. This technique is promising for pediatric imaging because it is portable, quick to perform, relatively low cost and involves no ionizing radiation. Acoustic force radiation imaging and ultrasound elastography does not have any increased risks over conventional ultrasound imaging.

DETAILED DESCRIPTION:
This is a single site prospective cohort study that will compare ultrasound elastography to traditional ultrasound parameters in bone marrow transplant patients who are at risk for development of SOS.

* Primary objective: compare sensitivity and specificity of traditional ultrasound parameters and ultrasound elastography of the liver for detecting SOS in BMT patients.
* Secondary objectives: 1. compare sensitivity and specificity of traditional ultrasound parameters and ultrasound elastography of the liver for classifying SOS in BMT patients. 2. compare sensitivity and specificity of traditional ultrasound parameters and ultrasound elastography of the liver for predicting death in BMT patients with SOS (defined as death within 100 days of transplant).
* The validity and reliability of the primary and secondary measures when available. The validity of the measures will be determined by comparing to clinical gold standards of the diagnosis and classification of SOS

Data Collection Procedures

* Candidates for the study will be identified by the Hematology Oncology service when they are admitted for bone marrow transplant.
* A member of the study team will consent that patient and/or their parents once the patient has been identified.
* If the patient consents to the study, an initial limited abdominal ultrasound with Doppler and shear wave elastography will be performed less than one month prior to bone marrow transplant. Demographic and clinical variables will be collected from the chart at the time of initial ultrasound and after date of discharge. Lab value variables will be collected at the time of the initial ultrasound and during all subsequent ultrasounds. Only lab values that have changed since the prior ultrasound will be recorded.
* Multiple shear wave elastography measurements of the liver will be obtained during any post-transplant clinical abdominal ultrasound Data Analyses We will perform two-sided t-tests and nonparametric tests for categorical and continuous data, respectively. Additionally, we will perform a multivariate regression to determine which variables are significantly correlated to death and calculate an odds ratio for each of these variables. If a patient is missing any imaging or clinical data, then this patient will be excluded from those parts of the data analysis, but the rest of their data will still be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are admitted for BMT from the date of study approval until patient accrual is met.

Exclusion Criteria:

* BMT patients who do not end up undergoing transplant during that admission. BMT patients who do not receive any abdominal ultrasounds post transplantation BMT patients who do not consent to the study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Chan, MD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] McDonald GB, Hinds MS, Fisher LD, Schoch HG, Wolford JL, Banaji M, Hardin BJ, Shulman HM, Clift RA. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993 Feb 15;118(4):255-67. doi: 10.7326/0003-4819-118-4-199302150-00003. PMID 8420443
- [Background] Carreras E, Bertz H, Arcese W, Vernant JP, Tomas JF, Hagglund H, Bandini G, Esperou H, Russell J, de la Rubia J, Di Girolamo G, Demuynck H, Hartmann O, Clausen J, Ruutu T, Leblond V, Iriondo A, Bosi A, Ben-Bassat I, Koza V, Gratwohl A, Apperley JF. Incidence and outcome of hepatic veno-occlusive disease after blood or marrow transplantation: a prospective cohort study of the European Group for Blood and Marrow Transplantation. European Group for Blood and Marrow Transplantation Chronic Leukemia Working Party. Blood. 1998 Nov 15;92(10):3599-604. PMID 9808553
- [Background] Hommeyer SC, Teefey SA, Jacobson AF, Higano CS, Bianco JA, Colacurcio CJ, McDonald GB. Venocclusive disease of the liver: prospective study of US evaluation. Radiology. 1992 Sep;184(3):683-6. doi: 10.1148/radiology.184.3.1509050.
- [Background] Teefey SA, Brink JA, Borson RA, Middleton WD. Diagnosis of venoocclusive disease of the liver after bone marrow transplantation: value of duplex sonography. AJR Am J Roentgenol. 1995 Jun;164(6):1397-401. doi: 10.2214/ajr.164.6.7754881.
- [Background] Garcia-Criado A, Gilabert R, Salmeron JM, Nicolau C, Vilana R, Bianchi L, Bunesch L, Garcia-Valdecasas JC, Rimola A, Bru C. Significance of and contributing factors for a high resistive index on Doppler sonography of the hepatic artery immediately after surgery: prognostic implications for liver transplant recipients. AJR Am J Roentgenol. 2003 Sep;181(3):831-8. doi: 10.2214/ajr.181.3.1810831. PMID 12933490
- [Background] Nicolau C, Bru C, Carreras E, Bosch J, Bianchi L, Gilabert R, Vilana R. Sonographic diagnosis and hemodynamic correlation in veno-occlusive disease of the liver. J Ultrasound Med. 1993 Aug;12(8):437-40. doi: 10.7863/jum.1993.12.8.437. PMID 8411325
- [Background] Herbetko J, Grigg AP, Buckley AR, Phillips GL. Venoocclusive liver disease after bone marrow transplantation: findings at duplex sonography. AJR Am J Roentgenol. 1992 May;158(5):1001-5. doi: 10.2214/ajr.158.5.1566656.
- [Background] Bamber J, Cosgrove D, Dietrich CF, Fromageau J, Bojunga J, Calliada F, Cantisani V, Correas JM, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Gilja OH, Havre RF, Jenssen C, Klauser AS, Ohlinger R, Saftoiu A, Schaefer F, Sporea I, Piscaglia F. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 1: Basic principles and technology. Ultraschall Med. 2013 Apr;34(2):169-84. doi: 10.1055/s-0033-1335205. Epub 2013 Apr 4. PMID 23558397
- [Background] Cosgrove D, Piscaglia F, Bamber J, Bojunga J, Correas JM, Gilja OH, Klauser AS, Sporea I, Calliada F, Cantisani V, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Fromageau J, Havre RF, Jenssen C, Ohlinger R, Saftoiu A, Schaefer F, Dietrich CF; EFSUMB. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 2: Clinical applications. Ultraschall Med. 2013 Jun;34(3):238-53. doi: 10.1055/s-0033-1335375. Epub 2013 Apr 19. PMID 23605169
- [Background] Shiina T, Nightingale KR, Palmeri ML, Hall TJ, Bamber JC, Barr RG, Castera L, Choi BI, Chou YH, Cosgrove D, Dietrich CF, Ding H, Amy D, Farrokh A, Ferraioli G, Filice C, Friedrich-Rust M, Nakashima K, Schafer F, Sporea I, Suzuki S, Wilson S, Kudo M. WFUMB guidelines and recommendations for clinical use of ultrasound elastography: Part 1: basic principles and terminology. Ultrasound Med Biol. 2015 May;41(5):1126-47. doi: 10.1016/j.ultrasmedbio.2015.03.009. Epub 2015 Mar 21. PMID 25805059
- [Background] Stenzel M, Mentzel HJ. Ultrasound elastography and contrast-enhanced ultrasound in infants, children and adolescents. Eur J Radiol. 2014 Sep;83(9):1560-9. doi: 10.1016/j.ejrad.2014.06.007. Epub 2014 Jun 28. PMID 25022978
- [Background] Ferraioli G, Filice C, Castera L, Choi BI, Sporea I, Wilson SR, Cosgrove D, Dietrich CF, Amy D, Bamber JC, Barr R, Chou YH, Ding H, Farrokh A, Friedrich-Rust M, Hall TJ, Nakashima K, Nightingale KR, Palmeri ML, Schafer F, Shiina T, Suzuki S, Kudo M. WFUMB guidelines and recommendations for clinical use of ultrasound elastography: Part 3: liver. Ultrasound Med Biol. 2015 May;41(5):1161-79. doi: 10.1016/j.ultrasmedbio.2015.03.007. Epub 2015 Mar 20. PMID 25800942
- [Background] Sugitani M, Fujita Y, Yumoto Y, Fukushima K, Takeuchi T, Shimokawa M, Kato K. A new method for measurement of placental elasticity: acoustic radiation force impulse imaging. Placenta. 2013 Nov;34(11):1009-13. doi: 10.1016/j.placenta.2013.08.014. Epub 2013 Sep 4. PMID 24075540
- [Background] Kutty SS, Peng Q, Danford DA, Fletcher SE, Perry D, Talmon GA, Scott C, Kugler JD, Duncan KF, Quiros-Tejeira RE, Kutty S; Liver Adult-Pediatric-Congenital-Heart-Disease Dysfunction Study (LADS) Group. Increased hepatic stiffness as consequence of high hepatic afterload in the Fontan circulation: a vascular Doppler and elastography study. Hepatology. 2014 Jan;59(1):251-60. doi: 10.1002/hep.26631. Epub 2013 Nov 19. PMID 23913702
- [Background] Leschied JR, Dillman JR, Bilhartz J, Heider A, Smith EA, Lopez MJ. Shear wave elastography helps differentiate biliary atresia from other neonatal/infantile liver diseases. Pediatr Radiol. 2015 Mar;45(3):366-75. doi: 10.1007/s00247-014-3149-z. Epub 2014 Sep 20. PMID 25238807
- [Background] Ozmen E, Adaletli I, Kayadibi Y, Emre S, Kilic F, Dervisoglu S, Kurugoglu S, Senyuz OF. The impact of share wave elastography in differentiation of hepatic hemangioma from malignant liver tumors in pediatric population. Eur J Radiol. 2014 Sep;83(9):1691-7. doi: 10.1016/j.ejrad.2014.06.002. Epub 2014 Jun 13. PMID 25012068
- [Background] Lin P, Chen M, Liu B, Wang S, Li X. Diagnostic performance of shear wave elastography in the identification of malignant thyroid nodules: a meta-analysis. Eur Radiol. 2014 Nov;24(11):2729-38. doi: 10.1007/s00330-014-3320-9. Epub 2014 Aug 12. PMID 25113648
- [Background] Liu B, Liang J, Zheng Y, Xie X, Huang G, Zhou L, Wang W, Lu M. Two-dimensional shear wave elastography as promising diagnostic tool for predicting malignant thyroid nodules: a prospective single-centre experience. Eur Radiol. 2015 Mar;25(3):624-34. doi: 10.1007/s00330-014-3455-8. Epub 2014 Oct 9. PMID 25298171
- [Background] Lacourpaille L, Hug F, Guevel A, Pereon Y, Magot A, Hogrel JY, Nordez A. Non-invasive assessment of muscle stiffness in patients with Duchenne muscular dystrophy. Muscle Nerve. 2015 Feb;51(2):284-6. doi: 10.1002/mus.24445. Epub 2014 Dec 23. PMID 25187068
- [Result] Reddivalla N, Robinson AL, Reid KJ, Radhi MA, Dalal J, Opfer EK, Chan SS. Using liver elastography to diagnose sinusoidal obstruction syndrome in pediatric patients undergoing hematopoetic stem cell transplant. Bone Marrow Transplant. 2020 Mar;55(3):523-530. doi: 10.1038/s41409-017-0064-6. Epub 2018 Jan 15. PMID 29335626

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shear Wave Ultrasound Elastography
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Shear Wave Ultrasound Elastography
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of US for VOD/SOS
Time Frame: within 100 days of bone marrow transplant
Measure: Number; unit: percentage of participants
Arm/Group | Shear Wave Ultrasound Elastography
Number analyzed (Participants) | 45
percentage of participants
  Sensitivity | 80
  Specificity | 93

2. Secondary Outcome: Severity of SOS
Description: death as noted in medical record
Time Frame: within 100 days of bone marrow transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Shear Wave Ultrasound Elastography
Number analyzed (Participants) | 45
Participants | 2

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Shear Wave Ultrasound Elastography
All-Cause Mortality (participants affected / at risk) | 11/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT02483481/Prot_SAP_000.pdf